CLINICAL TRIAL: NCT02287636
Title: Clinical Evaluation of PET-MRI Versus PET-CT in Pediatric Oncology Patients
Brief Title: PET/MRI and PET/CT in Diagnosing Younger Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE1Z13; NCI-2014-00828 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1Z13; CASE 1Z13 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-11-11 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (fludeoxyglucose F 18 PET/CT and PET/MRI) (Experimental): Patients undergo fludeoxyglucose F 18 PET/CT followed by PET/MRI.
  Interventions: Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography; Procedure: magnetic resonance imaging

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo fludeoxyglucose F 18 PET/CT
  Other Names: tomography, computed
Procedure: positron emission tomography — Undergo PET/MRI
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: magnetic resonance imaging — Undergo PET/MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
This pilot clinical trial studies how well positron emission tomography (PET)/magnetic resonance imaging (MRI) works compared to PET/computed tomography (CT) in diagnosing younger patients with cancer. PET/MRI and PET/CT are procedures that combine the pictures from a PET scan and an MRI scan or a CT scan. The PET and MRI scans or PET and CT scans are done at the same time with the same machine. The combined scans give more detailed pictures of areas inside the body than either scan gives by itself. It is not yet known whether PET/MRI works better than PET/CT in diagnosing younger patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the diagnostic accuracy of PET/MRI as compared to the standard of reference PET/CT in lesion detection and lesion characterization.

SECONDARY OBJECTIVES:

I. Obtain quantitative measurements in various body regions of standardized uptake values (SUV) in normal tissue and foci of pathologic tracer uptake in PET/MRI of pediatric patients with oncologic disease using various magnetic resonance attenuation correction (MRAC) methods and compare those to respective SUV based on CT attenuation correction.

II. Assess the potential for radiation dose reduction with PET/MRI when eliminating CT radiation dose.

III. Assess time efforts and workflow improvement with PET/MRI compared to sequential PET/CT plus MRI.

OUTLINE:

Patients undergo fludeoxyglucose F 18 PET/CT followed by PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred by their physician for clinically indicated diagnostic fludeoxyglucose F 18 (18F-FDG) PET/CT (with or without clinically indicated diagnostic MRI)
* Subjects with malignancies including hematologic disorders
* Subjects NOT requiring sedation or anesthesia
* Stable physical medical conditions (patients conscious and comfortable, scheduled for an elective diagnostic imaging)

Exclusion Criteria:

* Subjects who are unable or unwilling to give their assent to both examinations if > 7 years old
* Subjects requiring general anesthesia or sedation in order to undergo PET/CT or MRI
* Subjects unable to undergo magnetic resonance (MR) scanning due to exclusion by University Hospitals-Case Medical Center restriction policies for Magnetic Resonance Imaging (UHCMC MRI restriction policies) as mentioned in the standard UHCMC MRI informed consent form
* Previously known allergies against MRI contrast agents (exclusion criterion only for contrast enhanced MRI)
* Pregnant or breast feeding subjects, as determined by standard questionnaire administered prior to scanning

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bangert, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  0-9 years | 2
  10-19 years | 11
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 7
  Gender: Male | 5
  Gender: Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 4
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of PET/MRI
Description: Evaluation of the PET/MR imaging platform will be based on the ability to detect lesions. Evaluation of each lesion will be recorded using the following 5 point rating scale: 1=benign, 2=probably benign, 3=indeterminate, 4=probably malignant, 5=malignant. A Wilcoxon (Mann-Whitney) rank-sum test and two-sided z-test will be used to compare diagnostic accuracy of PET/MRI with PET/CT.
Time Frame: 1 day
Population: Sincere efforts were made to gather and report the data, however, no data is available for the study as PI has left institution long ago and not accessible.
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

2. Primary Outcome: Diagnostic Accuracy of PET/CT
Description: Evaluation of the PET/CT imaging platform will be based on the ability to detect lesions. Evaluation of each lesion will be recorded using the following 5 point rating scale: 1=benign, 2=probably benign, 3=indeterminate, 4=probably malignant, 5=malignant. A Wilcoxon (Mann-Whitney) rank-sum test and two-sided z-test will be used to compare diagnostic accuracy of PET/CT with PET/MRI.
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

3. Secondary Outcome: SUVs Using PET/MRI
Description: The means and standard deviations of SUVs will be obtained and compared between PET/MRI and PET/CT using a two-sided two-sample t-test.
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

4. Secondary Outcome: SUVs Using PET/CT
Description: as for outcome 3
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

5. Secondary Outcome: Radiation Dose Reduction Associated With PET/MRI
Description: Tabulations of summary statistics, graphical presentations, and statistical analyses will be performed. Statistical tests will use a 0.10 significance level and will be 2-sided unless otherwise noted. Confidence intervals, both individual and simultaneous, will be at 90% confidence level unless stated otherwise.
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time Effort Associated With the PET/MRI
Description: as for outcome 5
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At time of scan
Description: No adverse events were documented for this study
Arm/Group | Diagnostic (Fludeoxyglucose F 18 PET/CT and PET/MRI)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Sincere efforts were made to gather and report the data, however, no data is available for the study as PI has left institution long ago and not accessible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes